CLINICAL TRIAL: NCT04818931
Title: Does a Preoperative Prophylactic Antibiotic Reduce Surgical Site Infection Following Wire-localized Lumpectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2018-4107
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cefazolin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antibiotics (Experimental): Cefazolin 2 g or clindamycin 900 mg in case of penicillin allergy
  Interventions: Drug: Cefazolin Injection
- No antibiotics (No Intervention)

INTERVENTIONS:
Drug: Cefazolin Injection — cefazolin 2 g or clindamycin 900 mg in case of penicillin allergy
  Arms: Antibiotics

SUMMARY:
Background: Data on the benefits of preoperative prophylactic antibiotics for breast surgery are conflicting and there is no guideline for their use for wire-localized lumpectomy. The aims of this study were to determine whether a single dose of pre-operative antibiotic reduces surgical site infection (SSI) for wire-localized lumpectomy and to identify risk factors for SSI.

Methods: This was a prospective randomized trial carried out from April 2018 to June 2019 at the "Centre des Maladies du Sein du CHU de Québec - Université Laval", a tertiary center specialized in breast surgery. After informed consent, patients who underwent wire-localized lumpectomy were randomized to receive or not a pre-operative single dose of prophylactic antibiotic (cefazolin 2 g or clindamycin 900 mg in case of penicillin allergy). Data regarding demographics, comorbidities, perioperative details, and SSI were analyzed. SSI was considered if: 1) patient had positive wound cultures; or 2) required abscess drainage; or 3) received antibiotic treatment for breast symptoms (e.g., swelling, erythema, congestion) within 30 days after operation, in the absence of wound culture or in the presence of negative results. The patients and the investigator responsible for data collection were blind to grouping. All patients were called 30 days after surgery to be sure that they did not consult at another hospital for surgical wound infection.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* female
* scheduled for a wire-localized lumpectomy

Exclusion Criteria:

* pregnant or breastfeeding women
* incapacity to give informed consent
* preoperative breast infection
* patients known to be colonized with MRSA
* immunocompromised patients
* preoperative antibiotic prophylaxis needed for any concomitant condition.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2018-04-07 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with surgical site infection in each group | within 30 days after operation
  1) patient had positive wound cultures; or 2) required abscess drainage; or 3) received antibiotic treatment for breast symptoms (e.g., swelling, erythema, congestion)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Québec - Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Giguere GB, Poirier B, Provencher L, Boudreau D, Leblanc D, Poirier E, Hogue JC, Morin C, Desbiens C. Do Preoperative Prophylactic Antibiotics Reduce Surgical Site Infection Following Wire-Localized Lumpectomy? A Single-Blind Randomized Clinical Trial. Ann Surg Oncol. 2022 Apr;29(4):2202-2208. doi: 10.1245/s10434-021-11031-9. Epub 2021 Nov 25. PMID 34825283